CLINICAL TRIAL: NCT05972252
Title: A Feasibility Study to Evaluate the Safety and Efficacy of the Cerebrovascular Interventional Procedural Control System in Treatment of Acute Ischemic Stroke
Brief Title: First-in-man Study of the Cerebrovascular Interventional Procedural Control System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangzhou Dinova Neuroscience Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNS-CIPCS-01
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Patients with acute ischemic stroke will receive interventional procedure by the Cerebrovascular Interventional Procedural Control System.
  Interventions: Device: Cerebrovascular Interventional Procedural Control System

INTERVENTIONS:
Device: Cerebrovascular Interventional Procedural Control System — The Cerebrovascular Interventional Procedural Control System is intended for use in the remote delivery and manipulation of guidewires and rapid deliver stent catheters, and remote manipulation of guide catheters during cerebrovascular intervention procedures.

SUMMARY:
The objective of this study the first human use of a new device in treatment of acute ischemic stroke, which to evaluate the feasibility, safety, and efficacy of the Cerebrovascular Interventional Procedural Control System.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80.
2. Diagnosed with acute ischemic stroke.
3. Arterial occlusion in the anterior cerebral circulation that was confirmed by CTA or MRA.
4. Subject could be treated intraarterially within 8 hours after symptom onset.
5. Prestroke Modified Rankin Score ≤ 1.
6. National Institutes of Health Stroke Scale (NIHSS) ≥6 and ≤20.
7. Patients or their legally authorised representatives provided signed, informed consent.

Exclusion Criteria:

1. NCCT ASPECT score <6，or the infarct volume exceeded 1/3 of the middle cerebral artery blood supply area.
2. CT/MR Showed midline shift or cerebral hernia, and ventricle occupying effect. Intracranial hemorrhage. CTA/MRA shows carotid artery dissection, severe stenosis, or complete occlusion, which requiring carotid stent implantation during thrombectomy; Bilateral acute stroke or multiple intracranial large vessel occlusion.
3. Females who are pregnant or lactating.
4. Severe allergy to contrast agents, nickel-titanium metal or its alloys.
5. Drug-resistant hypertension (defined as sustained systolic blood pressure >185mmHg or diastolic blood pressure >110mmHg).
6. Hemorrhagic tendency (including but not limited to platelet <100*109/L, heparin treatment within 48 hours with APTT ≥35s, taking warfarin with an INR > 1.7).
7. Surgery or biopsy of parenchymal organs within the last 1 month
8. Any active or recent bleeding (gastrointestinal, urinary, etc.) within the last 1 month
9. Undergoing hemodialysis or peritoneal dialysis; exist of severe renal insufficiency (serum creatinine >220umol/L or 2.5mg/dl)
10. Previous intracranial hemorrhage, subarachnoid hemorrhage, brain tumor.
11. Life expectancy of less than 1 year.
12. Enrollment in another clinical trial evaluating other devices or drugs during the same period.
13. Abnormalities or diseases that the investigator considers to be excluded from the study's coverage.

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Good Neurological Outcome | 90±7 Days post-treatment
  Good clinical outcome is defined as an modified Rankin Scale (mRS) score of 0-2 at 90 days.
  mRS 0-2 indicates functional independence 0 - No symptoms.
Technical Success | Immediately post-treatment
  Using Cerebrovascular Interventional Procedural Control System successfully complete the catheters in placement, thrombectomy stent release, and thrombectomy system recovery, without manual conversion.

SECONDARY OUTCOMES:
Successful Revascularization | Immediately post-treatment
  Achieving mTICI ≥2b in the target vessel within 3 passes of the cerebrovascular interventional procedural control system without the use of rescue therapy.
Time from Groin Puncture to Reperfusion | Immediately post-treatment
  Time from groin puncture to achievement of mTICI ≥2b
Successful Recanalization Rate | Immediately post-treatment
  Achieving mTICI ≥2b in the target vessel within 1 passes of the Cerebrovascular Interventional Procedural Control System without the use of rescue therapy.
Radiation Exposure | Immediately post-treatment
  Total fluoroscopy dose utilized during the procedure as recorded by the DSA Imaging System.
Symptomatic Intracranial Hemorrhage | 36 hours post-treatment
  Symptomatic hemorrhage within 24 hours of procedure. Symptomatic hemorrhages is defined as any parenchymal hematoma 1 (PH1), parenchymal hematoma 2 (PH2), intraparenchymal hemorrhage remote from the ischemic field (RIH), intraventricular hemorrhage (IVH), and subarachnoid hemorrhage (SAH) associated with a worsening of National Institutes of Health Stroke Scale (NIHSS) ≥ 4 within 24hrs.
Device-related Serious Adverse Events (SAEs) | Through 90 days
  Any serious adverse events related to the device, such as vessel perforation, vessel dissection, vessel rupture, and severe spasm.
All-cause Mortality at 90 days | Through 90 days
  Rate of mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided